CLINICAL TRIAL: NCT00653133
Title: Multicenter Continuous Peripheral Nerve Block Surveillance Study Comparing Ultrasound Guided Catheter Placement to Non Ultrasound Guided Catheter Placement Techniques
Brief Title: Multicenter Continuous Peripheral Nerve Block Surveillance Study
Acronym: cpnb
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Halyard Health (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: iflocpnb2007
Record Dates: First submitted 2008-03-28; First posted 2008-04-04 (Estimated); Results first posted 2013-08-19 (Estimated); Last update posted 2018-10-02 (Actual); Status verified 2014-12

CONDITIONS: Postoperative Pain
Keywords: ultrasonography; peripheral nerve block; peripheral nerve stimulation
MeSH Terms: conditions — Pain, Postoperative | interventions — Ultrasonography

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- USPNB (Active Comparator): Ultrasound imaging guided peripheral nerve block
  Interventions: Device: Ultrasound imaging
- NSPNB (Active Comparator): Peripheral nerve stimulator guided peripheral nerve block catheter placement for continuous infusion of local anesthetic
  Interventions: Device: Peripheral nerve stimulator

INTERVENTIONS:
Device: Ultrasound imaging — Ultrasound guided techniques for placement of peripheral nerve block catheters for continuous infusion of local anesthetic
  Arms: USPNB
Device: Peripheral nerve stimulator — either stimulating needle or stimulating catheter used for placement of catheter for continuous infusion of local anesthetic
  Arms: NSPNB

SUMMARY:
This two tiered study is a multi-center, open label, surveillance study of the use of continuous nerve blocks with the ON-Q® C-bloc and either nerve stimulator or ultrasound guided continuous nerve block techniques. This study was developed to investigate specific aspects of complication rates related to continuous nerve block techniques in patients undergoing orthopedic surgical procedures.

DETAILED DESCRIPTION:
Continuous peripheral nerve block techniques require the placement of catheters near target peripheral nerves. The placement of these catheters is guided by either ultrasound visualization, nerve stimulation or a combination of the two.

This surveillance study was designed to look at the rates of catheter placement related complications with the two techniques.

ELIGIBILITY:
Inclusion Criteria:

* Patients having elective orthopedic surgery who are candidates for CPNB as part of their management program for postoperative pain
* Age >18
* Able to give consent

Exclusion Criteria:

* Morbid obesity (BMI> 40)
* Uncooperative or having psychological or linguistic difficulties
* Previous damage to the nerve or plexus
* Significant comorbidities which the primary investigator feels would limit the quality and collection of data
* Allergy to local anesthetic agents including ropivacaine, bupivacaine and lidocaine

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1821 (Actual)
Dates: Start 2007-05; Primary Completion 2009-03 (Actual); Study Completion 2009-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Joe Rodrigo, MD, Principal Investigator — Roper Hospital, Charleston, SC
Locations (16):
- United States (16):
  - Arizona Joint and Spine, Chandler, Arizona
  - Santa Clara Valley Medical Center, San Jose, California
  - Avista Adventist Hospital, Louisville, Colorado
  - Kennestone Hospital, Atlanta, Georgia
  - The Medical Center of Bowling Green, Bowling Green, Kentucky
  - Caritas Good Samaritan, Stoughton, Massachusetts
  - Wesley Medical Center, Hattiesburg, Mississippi
  - DesPeres Hospital, St Louis, Missouri
  - St. Vincents Catholic Medical Center, New York, New York
  - Charlotte Medical Center, Charlotte, North Carolina
  - Miami Valley Hospital, Dayton, Ohio
  - Bailey Medical Center, Owasso, Oklahoma
  - Roper Hospital, Charleston, South Carolina
  - Memorial Herman Hospital, Houston, Texas
  - Titus Regional Medical Center, Mount Pleasant, Texas
  - Virginia Commonwealth University, Richmond, Virginia

RESULTS

PARTICIPANT FLOW:
Groups:
- NSPNB: Stimulator guided nerve block
Period: Overall Study
Arm/Group | USPNB | NSPNB
Started | 1324 | 497
Completed | 1324 | 497
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | USPNB | NSPNB | Total
Number analyzed (Participants) | 1324 | 497 | 1821
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 12 | 0 | 12
  Between 18 and 65 years | 843 | 306 | 1149
  >=65 years | 469 | 191 | 660
Age, Continuous [Mean (Standard Deviation); unit: years] | 57.1 (16.4) | 57.7 (17.2) | 57.3 (16.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 649 | 214 | 863
  Male | 675 | 283 | 958
Region of Enrollment [Number; unit: participants]
  United States | 1324 | 497 | 1821

OUTCOME MEASURES:

1. Primary Outcome: Complications of Peripheral Nerve Block
Description: Adverse events related to performance of peripheral nerve catheter placement for continuous infusion of local anesthetic
Time Frame: Preoperative through 3 days post operative
Population: Intent to treat (ITT)
Measure: Number; unit: participants
Groups:
- NSPNB: Nerve Stimulator guided peripheral nerve block
Arm/Group | USPNB | NSPNB
Number analyzed (Participants) | 1324 | 497
participants | 7 | 14
Statistical Analysis 1: Comparison: USPNB vs NSPNB; Null hypothesis: There is no difference in reported complications associated with the placement of continuous peripheral nerve block catheters between ultrasound imaging guided placement and nerve stimulator guided placement; Test type: Superiority or Other; p < 0.05, t-test, 2 sided

ADVERSE EVENTS:
Time Frame: 7 days postoperative
Arm/Group | USPNB | NSPNB
Serious Adverse Events (participants affected / at risk) | 0/1324 | 0/497
Other Adverse Events (participants affected / at risk) | 7/1324 | 14/497
OTHER ADVERSE EVENTS (reported when occurring in more than 0.1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | USPNB (N=1324) | NSPNB (N=497)
VASCULAR PUNCTURE (Vascular disorders) | 4 (4) | 8 (8)
Infection (Infections and infestations) | 2 (2) | 2 (2) — CATHETER SITE LOCAL INFECTION/INFLAMMATION
motor block (Nervous system disorders) | 1 (1) | 4 (4)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No